CLINICAL TRIAL: NCT00178399
Title: A Pilot Study For Using Radiosurgery On Limited Metastases
Brief Title: A Study For Using Radiosurgery On Limited Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Michael Milano, MD,PhD, Associate Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: URCC 9700
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2018-10-11 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Neoplasms, Metastatic
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic body radiation therapy (Experimental)
  Interventions: Procedure: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Procedure: Stereotactic Body Radiation Therapy

SUMMARY:
The standard therapy in cases such as yours is surgery, radiation therapy, chemotherapy or hormonal therapy alone or in combination. The main purpose of this study is to evaluate whether radiosurgery alone affects your quality and length of life. A second purpose of this study is to determine if the levels of special types of protein (called cytokines) found in the blood are related to your quality of life during your course of treatment and follow-up.

DETAILED DESCRIPTION:
In this research study high dose stereotactic body radiation therapy will be directed at the site of metastasis. This treatment will be given once a day, 5 times a week (Monday through Friday) for one to four weeks depending on the location and size of the disease to be treated. Blood for the cytokine tests will be drawn before your therapy starts, weekly during therapy and at the follow-up visits as stated in the next paragraphs. Two to four tablespoons of blood will be removed each time.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years

KPS ≥ 70

Palliative: Disease most likely to be life limiting, is definable, and treatable to a sterilizing dose according to protocol criteria.

The size of the lesion must be such that it can be safely treated to sterilizing radiation doses according to the rules in the protocol

Previously treated lesions are not eligible unless the prescribed dose can be safely delivered. Previously enrolled patients can be retreated to new lesions if they still meet protocol requirements.

Informed consent must be obtained.

Pregnancy test must be negative for women of child bearing potential.

Out of state patients are eligible, if communication with the referring physicians is expected to be adequate to address the primary aim. The secondary aim (blood cytokines) is optional for out-of-state patients.

Exclusion Criteria:

Technical inability to achieve required dose based on safe dose constraints required for radiosurgery

Women who are pregnant or nursing..

Failure to meet inclusion requirements

Contraindications to radiation.

Patient should not be eligible for primary disease specific radiosurgical protocols

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2001-04 (Actual); Primary Completion 2007-03-15 (Actual); Study Completion 2007-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Milano, MD PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Department of Radiation Oncology, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Stereotactic Body Radiation Therapy: Stereotactic Body Radiation Therapy
Period: Overall Study
Arm/Group | Stereotactic Body Radiation Therapy
Started | 128
Completed | 115
Not Completed | 13
Not completed — Physician Decision | 4
Not completed — Withdrawal by Subject | 8
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 128
Age, Continuous [Median (Full Range); unit: years] | 60 [40 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 64
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 128

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Curatively Treated Patients With Progression-free Survival
Description: Curatively treated patients were those with metastatic disease confined to the thorax and or with total metastases limited to five total lesions.
Time Frame: 24 months
Population: Only curative patients were included in this analysis
Measure: Number; unit: percentage of participants
Groups:
- Stereotactic Body Radiation Therapy: Subjects received Stereotactic Body Radiation Therapy
Arm/Group | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 30
percentage of participants | 16

2. Primary Outcome: Percentage of Palliatively Treated Patients With Progression-free Survival
Description: Palliatively treated patients were those with more extensive disease wherein lung metastasis were considered the most life limiting component of their disease.
Time Frame: 24 months
Population: Only palliative patients were included in this analysis
Measure: Number; unit: percentage of participants
Arm/Group | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 19
percentage of participants | 38

3. Secondary Outcome: Quality of Life and Correlation With Pro-apoptotic, Inflammatory, and Anabolic Cytokine Profiles
Description: Correlation of data from QOL questionnaires and blood markers.
Time Frame: 30 months from date of registration.
Population: No data was collected for this outcome measure.
Arm/Group | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 0

4. Secondary Outcome: Analyze Impact of Disease Bulk and Number of Sites Involved.
Description: Analysis or response and progression.
Time Frame: From the date of radiation therapy treatment to the date of first failure or last follow-up, assessed up to 10 years
Population: No data was collected for this outcome measure.
Arm/Group | Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Stereotactic Body Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 123/128
Serious Adverse Events (participants affected / at risk) | 0/128
Other Adverse Events (participants affected / at risk) | 24/128
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stereotactic Body Radiation Therapy (N=128)
Pneumonitis/Pulmonary Infiltrates (Respiratory, thoracic and mediastinal disorders) | 20
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 2
Pericardial effusion (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes